CLINICAL TRIAL: NCT02752516
Title: Phase I Additional Study of Tolerance and Pharmacokinetics of Anlotinib in Patients With Advanced Solid Tumors
Brief Title: A Phase I Additional Study of Anlotinib on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-I-07
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib QD po. and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
A Phase I Additional Study of Anlotinib on Tolerance and Pharmacokinetics.To further study the pharmacokinetic characteristics of Anlotinib in the human body, recommend a reasonable regimen for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Advanced solid tumors except the digestive tract tumors,at least one measurable lesion (by RECIST1.1)
* Lack of the standard treatment or treatment failure
* 18-65 years,ECOG PS:0-1,Life expectancy of more than 3 months
* 30 Days or more from the last cytotoxic therapy
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients who are used by anlotinib
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Brain metastases patients with symptoms or symptoms controlled < 3 months
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  2. Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥480ms) and patients with Grade 1 or higher congestive heart failure (NYHA Classification);
  3. Patients with active or unable to control serious infections;
  4. Patients with cirrhosis, decompensated liver disease, or active hepatitis;
  5. Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L)
  6. Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed
* Patients with non-healing wounds or fractures
* Patients with any CTC AE Grade 1 or higher bleeding events occurred in the lungs or any CTC AE Grade 2 or higher bleeding events occurred within 4 weeks prior to assignment;Patients with any physical signs of bleeding diathesis or receiving thrombolysis and anticoagulation
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* Patients participated in other anticancer drug clinical trials within 4 weeks
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of Anlotinib (in whole blood):Peak Plasma Concentration(Cmax) | up to 18 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak Plasma Concentration(Cmax),Cmax in ng/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H72/H120/H168/H240（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D7/D10/D14/D18/Before the next cycle（D means Day）.
Pharmacokinetics of Anlotinib (in whole blood):Peak time（Tmax） | up to 18 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak time（Tmax）,Tmax in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H72/H120/H168/H240(H means hour).In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D7/D10/D14/D18/Before the next cycle(D means Day).
Pharmacokinetics of Anlotinib (in whole blood):Half life（t1/2） | up to 18 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Half life（t1/2）,t1/2 in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H72/H120/H168/H240(H mans Hour).In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D7/D10/D14/D18/Before the next cycle(D means Day).
Pharmacokinetics of Anlotinib (in whole blood):Area under the plasma concentration versus time curve (AUC) | up to 18 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Area under the plasma concentration versus time curve (AUC), AUC in ng.h/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H72/H120/H168/H240(H means Hour).In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D7/D10/D14/D18/Before the next cycle(D means Day).
Pharmacokinetics of Anlotinib (in whole blood):Clearance（CL） | up to 18 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Clearance（CL）,CL in L/h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H72/H120/H168/H240(H means Hour).In the study of multiple-dose,full PK profiles will be obtained at D1/D4/D7/D10/D14/D18/Before the next cycle(D means Day).
Cumulative excretion of Anlotinib (in urine) | up to 10 Days(endpoint when the two consecutive time points of cumulative excretion <1%)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD(Disease progression) (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided